CLINICAL TRIAL: NCT02817581
Title: Validation of National Early Warning Score (NEWS) and Rapid Lactate Testing for Early Identification of High Risk Patients in the Emergency Department
Brief Title: NEWS and Rapid Lactate Testing for Early Identification of High Risk Patients in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Colin Graham, Professor, Chinese University of Hong Kong
Other Study IDs: CRE- 2016.236
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Triage Category 3 (Urgent)
Keywords: National Early Warning Score (NEWS); Lactate; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To validate the NEWS and rapid lactate testing for early identification of high risk [triage Category 3 (urgent)] patients in the Emergency Department.

To compare qSOFA and SIRS criteria in patients in the Emergency Department.

DETAILED DESCRIPTION:
Background:

Sepsis is a potentially life-threatening complication of an infection. Early identification and early intervention are two main elements in improving patient care.

Objectives:

1. To validate the NEWS and rapid lactate testing for early identification of high risk [triage Category 3 (urgent)] patients in the Emergency Department.
2. To compare qSOFA and SIRS criteria in patients in the Emergency Department.

Study design:

This is a prospective, cohort study. Patients aged 18 or above presenting to the ED triaged as Category 3 (urgent) will be recruited. The required data for calculating NEWS will be collected at triage and triage lactate level will be measured by point-of-care analyzer.

Outcomes:

The primary outcome is referral for intensive care unit (ICU) admission during the patient's ED stay. The secondary outcomes are length of stay in hospital (LOS), hospital admission, admission to ICU, length of ICU-free admission (defined as days alive outside the ICU from admission to day 30) 30-day mortality and time to processes-of-care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above who are triage category 3 in emergency department
* Presenting to emergency department between 9am and 4pm, Monday to Friday

Exclusion Criteria:

* Aged below 18 years
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or above who are triage category 3 presenting to Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 1255 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days after recruitment

SECONDARY OUTCOMES:
referral for intensive care unit (ICU) admission | 24 hr after recruitment
length of stay in hospital (LOS) | 30 days after recruitment
hospital admission | 30 days after recruitment
admission to ICU | 30 days after recruitment
length of ICU-free admission | 30 days after recruitment
time to processes-of-care | 24 hr after recruitment
  time to lactate measured, time to antibiotics admission, time to blood culture obtained, time to fluid resuscitation, time to vasopressor administration from ED arrival

CONTACTS AND LOCATIONS:
Overall Officials: Colin A Graham, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, NT, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes